CLINICAL TRIAL: NCT01219270
Title: Radiocontrast Media Induced Hyponatremia After Percutaneous Coronary Intervention: Observational Study
Brief Title: Radiocontrast Media Induced Hyponatremia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Gachon University Gil Medical Center IRB, Gachon University Gil Medical Center
Other Study IDs: Hyponatremia-GUGH
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Radiocontrast media,; hyponatremia
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GFR >= 60: MDRD eGFR 60 or more
- GFR <60: Under MDRD eGFR 60

SUMMARY:
Osmolality of contrast media can be resulted in translocational hyponatremia after percutaneous coronary intervention.

DETAILED DESCRIPTION:
Radiocontrast media after percutaneous coronary interventioncan lead to increased osmolaliry of plasma, which results in translocational hyponatremia.

The investigator will exam the incidence of hyponatremia after percutaneous coronary intervention, and will evaluate the underlying mechanism related to hyponatremia including translocational hyponatremia, or osmotic natriuresis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive contrast media during percutaneous coronary intervention

Exclusion Criteria:

* Patients who have sensitivity to contrast media.
* Liver cirrhosis
* Hypothyroidism
* SIADH
* Patients who receive IVIG or mannitol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who receive contrast media during percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-02 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of contrast media induced translocational hyponatremia | 01/10/2010-28/02/2011
  The will investigator evaluate how often translocational hyponatremia may develop after percutaneous coronary intervention.

SECONDARY OUTCOMES:
Renal function is affected by the incidence of translocational hyponatremia. | 01/10/2010-28/02/2011
  Reduced renal function and urine output contribute the development of contrast media induced translocational hyponatremia.

CONTACTS AND LOCATIONS:
Overall Officials: Sejoong Kim, MD, PhD, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Hospital, Incheon, South Korea

REFERENCES:
- [Background] Aronson D, Dragu RE, Nakhoul F, Hir J, Miller A, Boulos M, Zinder O, Green J, Mittleman MA, Markiewicz W. Hyponatremia as a complication of cardiac catheterization: a prospective study. Am J Kidney Dis. 2002 Nov;40(5):940-6. doi: 10.1053/ajkd.2002.36324. PMID 12407638